CLINICAL TRIAL: NCT04568226
Title: The Effect of Metacognition-based, Manualized Intervention on Fear of Cancer Recurrence: a Randomized Controlled Trial
Brief Title: The Effect of Metacognition-based, Manualized Intervention on Fear of Cancer Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Wendy Wing Tak Lam, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW19-183
Record Dates: First submitted 2020-09-22; First posted 2020-09-29 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Fear of Cancer Recurrence
Keywords: Fear of cancer recurrence; Metacognition; Cancer survivorship; Psychooncology; Breast cancer; Colorectal cancer; Gynecologic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: We will use a block randomization structure with randomly permuted block sizes of 2,4, and 6 to ensure a close balance of the numbers in each arm. Randomization (by a statistician) occurs prior to eligible patients attending the clinic to minimize opportunities for selection bias.
  We will also use a block randomization structure with randomly permuted block sizes of 4 and 8 to ensure an equal case allocation to each therapist.
  We will also use a block randomization structure with randomly permuted block sizes of 2,4, and 6 to ensure an equal case allocation to each dietitian.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, care provider, and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to ConquerFear or control arms.
  The participants are masked in terms of not knowing that one intervention (i.e. Conquer fear) is hypothesized to yield larger effects than the other (i.e. control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ConquerFear Intervention (Experimental): Participants in the ConquerFear intervention group will receive a manualized intervention, consisting of 6 therapist-led individual sessions.
  Interventions: Other: ConquerFear Intervention
- Basic Cancer Care (Active Comparator): Basic Cancer Care serves as an active comparator and is not developed specifically to target fear of cancer recurrence through modifying participants' cognitive beliefs. Participants in this arm will receive 6 individual sessions including 2 relaxation training sessions, 2 dietetic consultation sessions, and 2 exercise sessions, which will be led by a trained therapist, a registered dietitian, and an exercise physiologist, respectively.
  Interventions: Other: Active control: Basic Cancer Care

INTERVENTIONS:
Other: ConquerFear Intervention — ConquerFear is a manualized intervention, consists of six individual sessions over 10 weeks. The key goals of this intervention are the following: (1) teach strategies for controlling worry and excessive threat monitoring, (2) modify underlying unhelpful beliefs about worry, (3) develop appropriate monitoring and screening behaviours, (4) encourage acceptance of the uncertainty brought about by a cancer diagnosis, and (5) clarify values and encourage engagement in values-based goal setting (19). Each session will last 60-90 minutes and be delivered by a trained therapist. After each session, participants will be given home-based exercises to practice the skills learned in the sessions. With the uncertainty surrounding the COVID-19 pandemic, instead of face-to-face sessions only, a hybrid mode of intervention delivery will be used by offering participants the choice of face-to-face or online sessions.
  Arms: ConquerFear Intervention
Other: Active control: Basic Cancer Care — Basic Cancer Care intervention for the control arm was developed to help cancer survivors with health maintenance in long-term through providing comprehensive lifestyle guidance. The intervention incorporates relaxation training, dietary and physical fitness consultations with the key goals to (1) teach relaxation techniques, (2) offer personalized diet and physical activity advice, and (3) enhance survivors' perceived control over illness, thereby leading to better adjustment to cancer. Similar to the ConquerFear intervention, Basic Cancer Care intervention consists of 6 individual sessions over 10 weeks. Each session will last 60-90 minutes and be delivered by a trained therapist, a registered dietitian, and an exercise physiologist, respectively. A hybrid mode of intervention delivery will be also used by offering participants the choice of face-to-face or online sessions.
  Arms: Basic Cancer Care

SUMMARY:
The primary aim of this study is to assess the effect of ConquerFear, a metacognition-based manualized intervention on fear of cancer recurrence, using the randomized controlled trial approach, among Chinese patients newly diagnosed with curable cancer. This study aims to (1) test the direct effect of ConquerFear intervention on fear of cancer recurrence and on maladaptive metacognition, and (2) to test the indirect effect of ConquerFear intervention on fear of cancer recurrence through its effect on maladaptive metacognition.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted to test the effect of a metacognition-based manualized intervention on fear of cancer recurrence among Chinese breast, gynecologic and colorectal cancer patients with high levels of fear of cancer recurrence.

The aims are to test:

1. the direct effect of ConquerFear intervention on fear of cancer recurrence,
2. the direct effect of ConquerFear intervention on maladaptive metacognition
3. the indirect effect of ConquerFear intervention on fear of cancer recurrence through its effect on maladaptive metacognition.

Primary hypothesis:

1. Participants in the ConquerFear intervention will show a greater reduction in fear of cancer recurrence compared to participants in the control group
2. Participants in the ConquerFear intervention will show a greater reduction in maladaptive metacognition than the control participants
3. There will be an indirect effect of ConquerFear intervention on fear of cancer recurrence through its effect on maladaptive metacognition.

ELIGIBILITY:
Inclusion Criteria:

1. Cantonese- or Mandarin-speaking Chinese patients recently diagnosed with non-metastatic breast cancer, gynecologic cancer, or colorectal cancer
2. had surgery as a primary treatment
3. have had completed hospital-based adjuvant treatments including radiotherapy and chemotherapy within the past 18 months
4. with the cut-off scored ≥ 13 on Severity, the subscale of Fear of cancer inventory
5. are able to read and write Chinese
6. are over the age of 18 years

Exclusion Criteria:

1. non-Chinese ethnicity
2. Patients diagnosed with metastatic cancer
3. with a current diagnosis of depression or psychosis
4. currently receiving psychological treatment
5. with language difficulties or intellectual disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-02-03 (Actual)

PRIMARY OUTCOMES:
Fear of cancer recurrence | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  The 42-items Fear of cancer recurrence inventory comprised of seven subscales will be used to assess the change of fear of cancer recurrence (FCR). Each item is rated on a 5-point Likert Scale with a total score ranging from 0 to 168. Higher scores indicate greater FCR. The subscale, Severity will be used as a screening tool for high level of FCR. A score of 13 or higher was optimal for screening.

SECONDARY OUTCOMES:
Metacognitions | Baseline, immediate post-intervention, 3months post-intervention, and 6months
  The 30-items Metacognitions questionnaire (MCQ-30) will be used to assess the change of metacognitive beliefs.Each item is rated on a 4-point Likert scale with a total score ranging from 30 to 120. High scores indicate a more maladaptive metacognitive style.
EORTC QLQ-C30 | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Quality of life (QoL) will be assessed by the EORTC QLQ-C30, in which incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease.
Self-efficacy | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Self-efficacy for managing chronic disease will be assessed using the Self-Efficacy for Managing Chronic Disease 6-item Scale.
Coping behavior | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Coping behavior will be assessed using the 28-item Chinese Brief COPE.
Experimental avoidance | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Experimental avoidance will be assessed using the Acceptance and action questionnaire.
Cognitive Attentional Syndrome | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Cognitive Attentional Syndrome (CAS) will be assessed using the Cognitive-attentional Syndrome questionnaire (CAS-1).
Intolerance of uncertainty | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Intolerance of uncertainty (IU) will be assessed using the 12-item Intolerance of uncertainty-12.
Psychological distress | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Psychological distress will be assessed using the Hospital Anxiety and Depression Scale (HADS). HADS is a 14-item measure of anxiety and depression widely used to assess cancer-related distress.
Cancer-related distress | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  The 22-item Chinese Impact of Events Scale-revised (CIES-R) will be used to assess cancer-related distress, which comprised three subscales: avoidance, intrusive thoughts and hyperarousal symptoms measured using 5-point Likert scales. Higher mean scores on each subscale indicate greater avoidance/intrusiveness/arousal.
Treatment expectancy | Baseline and immediate post-intervention
  Treatment expectancy will be assessed using the 6-item credibility/ expectancy questionnaire.
Therapeutic alliance | Immediate post-intervention
  The 12-item Working Alliance Inventory (WAI-SF)will be used to assess agreement on the therapy goal, patients' agreement with the therapist, and quality of the interpersonal bond. Both the participants and therapists will be asked to fill in the WAI-SF immediate post-intervention
Treatment satisfaction | Immediate post-intervention
  Treatment satisfaction will be assessed using the evaluation form. Participants will be asked to indicate their overall satisfaction with the intervention they have received.

OTHER OUTCOMES:
Demographic data | Baseline
  Demographic data including age, gender, marital status, education level, occupation and monthly family income will be assessed by self-reported questionnaire
Clinical data | Baseline, immediate post-intervention, 3months post-intervention, and 6months post-intervention
  Clinical data will be extracted from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wing Tak Lam, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (6):
- Hong Kong (6):
  - Queen Mary Hospital-Department of Surgery, Hong Kong
  - Kwong Wah Hospital-Breast Center, Hong Kong
  - Prince of Wales Hospital-Department of Surgery, Hong Kong
  - Queen Mary Hospital-Department of Obstetrics & Gynaecology, Hong Kong
  - The University of Hong Kong Jockey Club Institute of Cancer Care, Hong Kong
  - Tung Wah Hospital-Department of Surgery, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.

REFERENCES:
- [Background] Ng DWL, Foo CC, Ng SSM, Kwong A, Suen D, Chan M, Or A, Chun OK, Fielding BFS, Lam WWT. The role of metacognition and its indirect effect through cognitive attentional syndrome on fear of cancer recurrence trajectories: A longitudinal study. Psychooncology. 2020 Feb;29(2):271-279. doi: 10.1002/pon.5234. Epub 2019 Dec 23. PMID 31663187
- [Background] Ng DWL, Kwong A, Suen D, Chan M, Or A, Ng SS, Foo CC, Fielding BFS, Lam WWT. Fear of cancer recurrence among Chinese cancer survivors: Prevalence and associations with metacognition and neuroticism. Psychooncology. 2019 Jun;28(6):1243-1251. doi: 10.1002/pon.5073. Epub 2019 Apr 26. PMID 30932279
- [Background] Butow PN, Turner J, Gilchrist J, Sharpe L, Smith AB, Fardell JE, Tesson S, O'Connell R, Girgis A, Gebski VJ, Asher R, Mihalopoulos C, Bell ML, Zola KG, Beith J, Thewes B. Randomized Trial of ConquerFear: A Novel, Theoretically Based Psychosocial Intervention for Fear of Cancer Recurrence. J Clin Oncol. 2017 Dec 20;35(36):4066-4077. doi: 10.1200/JCO.2017.73.1257. Epub 2017 Nov 2. PMID 29095681
- [Derived] Ng DWL, Ng R, Guo C, Chan J, Fielding R, Tang JWC, Li WWY, Foo CC, Kwong A, Ng SS, Suen D, Fung S, Chun OK, Chan KKL, Chang ATY, Butow P, Lam WWT. ConquerFear-HK: A Randomized Controlled Trial of a Metacognition-Based, Manualized Intervention for Fear of Cancer Recurrence among Chinese Cancer Survivors. Psychother Psychosom. 2025 Aug 8:1-17. doi: 10.1159/000547888. Online ahead of print. PMID 40784346
- [Derived] Ng DWL, Fielding R, Tsang C, Ng C, Chan J, Or A, Kong IWM, Tang JWC, Li WWY, Chang ATY, Foo CC, Kwong A, Ng SS, Suen D, Chan M, Chun OK, Chan KKL, Butow PN, Lam WWT. Study protocol of ConquerFear-HK: a randomised controlled trial of a metacognition-based, manualised intervention for fear of cancer recurrence among Chinese cancer survivors. BMJ Open. 2023 Jan 20;13(1):e065075. doi: 10.1136/bmjopen-2022-065075. PMID 36669845